CLINICAL TRIAL: NCT03889548
Title: Influence of Resistance Training Experience on the Efficacy of Mental Imagery in Modulating Corticospinal Excitability and Inhibition: A Pilot Study
Brief Title: Influence of Resistance Training Experience and Mental Imagery on Corticospinal Excitability and Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Matt Stock, Assistant Professor, University of Central Florida
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 00000170
Record Dates: First submitted 2019-03-22; First posted 2019-03-26 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Resistance Training

STUDY DESIGN:
Intervention Model Description: Within-subjects design with mental imagery and control conditions performed in random order
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mental Imagery (Experimental)
  Interventions: Other: Mental Imagery
- Control (No Intervention)

INTERVENTIONS:
Other: Mental Imagery — Immediately after determination of the resting motor threshold and pre-test measurements, the TMS administrator will leave the room so as to be blinded to the treatment condition of the participant. At this time the participant will be given instructions regarding the mental imagery protocol from a separate investigator who will not be blinded to the condition. During the mental imagery protocol, participants will be instructed to close their eyes and imagine they are maximally contracting the muscles in their forearm and imagine that they are making their wrist flex and that they are pushing maximally against a hand grip in their hand. This will be a kinesthetic imagery task, in which they are urging their muscles to contract maximally.
  Arms: Mental Imagery

SUMMARY:
This study will utilize transcranial magnetic stimulation (TMS) to examine the effects of mental imagery in resistance-trained versus untrained men and women. In randomized order, each participant will perform a mental imagery task or a control condition as TMS is used to study corticospinal excitability.

DETAILED DESCRIPTION:
Kinesthetic mental imagery is a technique that has previously been utilized to modulate neural signaling to the limbs in the absence of any mechanical movement of the limb. Kinesthetic imagery tasks require an individual to imagine they are maximally contracting a target muscle group. Previous investigations have shown mental imagery tasks to increase maximal strength of the limb and even attenuate strength loss during periods of immobilization. Similarly, corticospinal excitability, which indicates the ease in which the cortex can stimulate muscular contraction, has also been shown to increase during mental imagery tasks. These adaptations have been attributed to the role of the cortex as a critical determinant of strength and the potent cortical stimulus posed by mental imagery.

Mental imagery and resistance training have both shown to provide a positive impact on muscle strength. However, the interplay between a mental imagery task and resistance training experience has yet to be fully investigated in terms of their impact on corticospinal excitability and inhibition. To our knowledge, no study has examined the effect of resistance training experience on corticospinal excitability and inhibition during a mental imagery task. Thus, the purpose of this study is to determine if resistance trained and untrained participants experience differences in corticospinal excitability and inhibition during kinesthetic mental imagery.

ELIGIBILITY:
Inclusion Criteria:

* Over the previous six months, participant has performed at least three resistance training sessions per week or
* Over the previous six months, participant has refrained from resistance training entirely.

Exclusion Criteria:

* Do not meet the resistance training experience requirements of either group
* Neuromuscular disease (e.g. Parkinson's, MS, ALS)
* Metabolic disease (e.g. diabetes, thyroid disorder, metabolic syndrome)
* Arthritis in the upper limbs (hands, arms, shoulders)
* Trouble using or controlling one's muscles
* History of cancer
* History of stroke
* History of heart attack
* Use of an assistive walking device or other mobility aids
* Physician mandated contraindication to exercise within the last 6 months
* Epilepsy or history of convulsions/seizures
* History of fainting or syncope
* History of head trauma that was diagnosed as concussion or was associated with loss of consciousness
* History of hearing problems or tinnitus
* Cochlear implants
* Implanted metal in the brain, skull, or elsewhere in the body
* Implanted neurotransmitter
* Cardiac pacemaker or intracardiac lines
* Medication infusion device
* Past problems with brain stimulation
* Past problems with MRI
* Use of muscle relaxants or benzodiazepines
* Allergy to rubbing alcohol
* Any other health related illnesses that would prohibit a participant from physical performance testing
* Lack of transportation to and from the laboratory
* Any permanent / non-removable jewelry or metal fixtures

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Corticospinal Excitability | Greater than or equal to 24 hours to 7 days between visits.
  Peak-to-peak amplitude of the motor evoked potential of the first dorsal interosseous at 130% of resting motor threshold

CONTACTS AND LOCATIONS:
Overall Officials: Matt S Stock, Ph.D., Principal Investigator — School of Kinesiology and Physical Therapy
Locations (1):
- Central Florida Research Park; Partnership 1 Building; UCF Neuromuscular Plasticity Laboratory, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Parsowith EJ, Stock MS, Girts RM, Beausejour JP, Alberto A, Carr JC, Harmon KK. The Influence of Resistance Training Experience on the Efficacy of Motor Imagery for Acutely Increasing Corticospinal Excitability. Brain Sci. 2023 Nov 25;13(12):1635. doi: 10.3390/brainsci13121635. PMID 38137083